CLINICAL TRIAL: NCT07338097
Title: Comparison of Bevacizumab and Aflibercept in Treatment of Diabetic Macular Edema
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Multan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Sana Javed, Principal Investigator, CMH Multan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIMS1
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Macular Edema (DME)
Keywords: Diabetic macular edema; Intravitreal injection; Anti vascular endothelial growth factor; Bevacizumab; Aflibercept; Visual acuity
MeSH Terms: interventions — aflibercept; Bevacizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Aflibercept (Experimental): Participants will receive intravitreal aflibercept administered as 2.0 mg injection, given monthly for two months.
  Interventions: Drug: Aflibercept (2.0 mg)
- Group Bevacizumab (Active Comparator): Participants will receive intravitreal bevacizumab administered as 1.25 mg injection, given monthly for two months
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Aflibercept (2.0 mg) — Intravitreal aflibercept 2.0 mg, administered once monthly for two consecutive months.
  Arms: Group Aflibercept
Drug: Bevacizumab — Intravitreal bevacizumab 1.25 mg, administered once monthly for two consecutive months.
  Arms: Group Bevacizumab

SUMMARY:
Diabetic macular edema is a frequent complication of long-standing diabetes mellitus in which fluid leaks into the central part of the retina (macula), leading to reduced vision. This randomized controlled trial will be conducted at Combined Military Hospital, Multan, to compare two commonly used intravitreal anti vascular endothelial growth factor medicines, aflibercept and bevacizumab, in adults aged 30 to 60 years with type 1 or type 2 diabetes mellitus for at least 5 years, central macular thickness of at least 300 micrometers on optical coherence tomography, and reduced baseline visual acuity (20/50 or worse). Eligible participants will be allocated in a 1:1 ratio to receive either intravitreal aflibercept 2.0 mg or intravitreal bevacizumab 1.25 mg, administered monthly for two months, with follow-up assessments at 1 and 2 months. The primary hypothesis is that aflibercept produces a greater average improvement in visual acuity than bevacizumab in this patient group. The primary outcome is the mean change in visual acuity measured as Early Treatment Diabetic Retinopathy Study letter score from baseline to 2 months. The secondary outcome is the mean change in central retinal thickness on optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or type 2 diabetes mellitus for ≥5 years
* Baseline visual acuity of 20/50 or worse
* Central macular thickness of ≥300 µm on OCT
* Age 30 to 60 years
* Either gender
* Provided voluntary consent for participation

Exclusion Criteria:

* History of prior treatment for DME: anti-VEGF, steroids, or laser.
* Active ocular infection or inflammation
* History of cardiac disease or stroke
* Women who are pregnant or breastfeeding
* Known allergy to Aflibercept or Bevacizumab
* Patient refusals to participate in the study

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-09-07 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Visual Acuity Letter Score | Baseline assessment before first injection and follow up evaluation at the end of 2 months after initiation of treatment.
  The primary outcome is the average change in visual acuity expressed as Early Treatment Diabetic Retinopathy Study (ETDRS) letter score, calculated by converting Snellen visual acuity measurements. The change is determined by subtracting baseline letter score from the letter score measured at follow up. This metric reflects functional improvement in vision.

SECONDARY OUTCOMES:
Mean Change in Central Retinal Thickness | Baseline assessment before first injection and follow up evaluation at the end of 2 months after initiation of treatment.
  The secondary outcome is the average change in central retinal thickness measured in micrometers using optical coherence tomography. The change is calculated by comparing baseline thickness with the value measured at follow up. This outcome reflects anatomical response of the macula to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Javed, Principal Investigator — CMH Institute of Medical Sciences
Locations (1):
- CMH Institute of Medical Sciences, Multan, Punjab Province, Pakistan